CLINICAL TRIAL: NCT04724486
Title: Effect of GnRH Agonist (Long Protocol) vs GnRH Antagonist (Flexible Protocol) on Oocyte Morphology During IVF/ICSI
Brief Title: Effect of GnRH Agonist vs GnRH Antagonist on Oocyte Morphology During IVF/ICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ph-CT-4301
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: In Vitro Fertilization; Intracytoplasmic Sperm Injection; Infertility
Keywords: GnRH Agonist; GnRH Antagonist; Oocyte morphology; Assisted reproduction technique; In Vitro Fertilization; Intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; cetrorelix; Menotropins; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agonist Group (Long protocol): (Active Comparator): The pituitary down-regulation in this group will be carried out using 0.05-0.1 mg of Triptorelin acetate subcutaneously (SC) once daily from the mid-luteal phase (day 21) of the menstrual cycle until the ovulation triggering day. When the suppressive effect is obtained, ovarian stimulation will commence with recombinant Follicle-Stimulating Hormone (r-FSH) or r-FSH + human Menopausal Gonadotropin (hMG) and the dose will be adjusted according to the ovarian response. Ovulation will be triggered by the administration of 10,000 IU of human Chorionic Gonadotropin (hCG) when at least three follicles become more than 16-17 mm. After 35±2 hours of ovulation triggering, the oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration. Then they will be prepared to undergo an Intracytoplasmic Sperm Injection (ICSI).
  Interventions: Drug: Triptorelin acetate; Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin; Drug: Human Chorionic Gonadotropin (hCG)
- Antagonist Group (Flexible protocol): (Experimental): The ovarian stimulation in this group will be started with recombinant Follicle-Stimulating Hormone (r-FSH) or r-FSH + human Menopausal Gonadotropin (hMG) on the third day of the menstrual cycle and the dose will be adjusted according to the ovarian response. Initiation of 0.25 mg of GnRH antagonist; Cetrorelix; will take place after detecting a leading follicle diameter ≥ 14 mm. GnRH antagonist administration will be continued till the day of ovulation triggering, which will be accomplished by given 10,000 IU of human Chorionic Gonadotropin (hCG) when at least three follicles become more than 16-17 mm. After 35±2 hours of ovulation triggering, the oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration. Then they will be prepared to undergo an Intracytoplasmic Sperm Injection (ICSI).
  Interventions: Drug: Cetrorelix; Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin; Drug: Human Chorionic Gonadotropin (hCG)

INTERVENTIONS:
Drug: Triptorelin acetate — 0.05-0.1 mg subcutaneously (SC) once daily from the mid-luteal phase (day 21) of the cycle until the day of ovulation triggering.
  Arms: Agonist Group (Long protocol):
Drug: Cetrorelix — 0.25 mg subcutaneously (SC) once daily starting from the day detecting a leading follicle diameter ≥ 14 mm until the day of ovulation triggering.
  Arms: Antagonist Group (Flexible protocol):
Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin — Dosage adjustment according to the ovarian response.
Drug: Human Chorionic Gonadotropin (hCG) — Ovulation will be triggered by the administration of 10,000 IU of human chorionic gonadotropin when at least three follicles become more than 16-17 mm.

SUMMARY:
Selection of developmentally competent oocytes enhances IVF efficiency. Usually, oocyte quality is determined based on its nuclear maturation and the presence of specific cytoplasmic and extracytoplasmic morphologic features. Gonadotropin-releasing hormone agonists (GnRH Agonists) and gonadotropin-releasing hormone antagonists (GnRH Antagonists) are used during controlled ovarian stimulation (COS) protocols in order to prevent premature luteinizing hormone (LH) surge and premature ovulation. However, GnRH receptors are also expressed in extra-pituitary tissues such as ovary, but it is still unknown whether the type of GnRH analogues used during COS could affect the oocyte morphology, especially with the limited and conflicted currently available data. Thus, we are conducting this prospective, non-randomised, open-label, clinical trial to compare the effects of two pituitary suppression regimens; GnRH Agonist-Long Protocol and GnRH Antagonist-Flexible Protocol on oocyte morphology during IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF/ICSI.
* Age: 18-39 years.
* Both ovaries present.

Exclusion Criteria:

* Age ≥ 40 years
* History of three or more previous IVF failures.
* Patients with hormonal disorders like hyperprolactinemia, thyroid disorders.
* Patients with Polycystic Ovarian Syndrome.
* Patients who previously undergo Unilateral Oophorectomy.
* Patients with chronic diseases: diabetes mellitus, cardiovascular diseases, liver diseases, kidney diseases.
* Patients with diseases may affect IVF outcomes: Endometriosis, uterine fibroids, Hydrosalpinx, Adenomyosis, autoimmune diseases,
* Cancer.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of oocyte dysmorphisms among the studied groups: | Before oocytes microinjection
  Before being subjected to ICSI, the oocytes from both groups will be morphologically analyzed under an inverted microscope; Nikon Eclipse Ti2; in order to detect cytoplasmic and extra-cytoplasmic dysmorphisms.

SECONDARY OUTCOMES:
Number of oocytes retrieved: | Immediately after oocyte retrieval (35±2 hours after hCG administration)
  The oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration 35±2 hours after hCG administration.
Number of Metaphase II Oocytes (MII): | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope.
Number of Metaphase I Oocytes (MI): | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope.
Number of Germinal Vesicle Oocytes (GV): | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope.
Number of Atretic Oocytes: | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope.
Maturation Rate%: | Within two hours after oocyte retrieval
  Maturation Rate is calculated by dividing the number of mature (MII) oocytes by the number of retrieved oocytes.
Fertilization Rate%: | 16-18 hours after microinjection
  Fertilization Rate is calculated by dividing the number of obtained zygote (2PN) by the number of injected oocytes.
Cleavage Rate%: | Day 2 after microinjection
  Cleavage rate is calculated by dividing the number of cleavaged embryos by the number of zygotes (2PN).
Embryo Quality: | Day of transfer (2 or 3 days after microinjection)
  Embryos are assessed using Nikon SMZ1500 stereoscope based on ESHRE criteria (2011).
High Quality Embryos rate%: | Day of transfer (2 or 3 days after microinjection)
  High Quality Embryos rate is calculated by dividing the number of high quality embryos (Grade I) by the total number of cleavaged embryos.
Biochemical Pregnancy Rate% (Per Embryo Transfer): | 2 weeks after embryo transfer
  Biochemical pregnancy is defined as a positive serum beta-hCG pregnancy test after 2 weeks of embryo transfer. The biochemical pregnancy rate is calculated by dividing the number of women who are biochemically pregnant by the number of women who have at least 1 embryo transferred.
Clinical Pregnancy Rate% (Per Embryo Transfer): | 3-4 weeks after embryo transfer
  Clinical pregnancy is defined as the presence of a gestational sac on ultrasound after 3-4 weeks of embryo transfer. The clinical pregnancy rate is calculated as by dividing the number of women who are clinically pregnant divided by the number of women who have at least 1 embryo transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Kadoura, B Pharm, MD, Principal Investigator — Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Abdul Hakim Nattouf, MD, PhD, Study Director — Professor at Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Marwan Alhalabi, MD, PhD, Study Director — Professor at Department of Embryology and Reproductive Medicine, Faculty of Medicine, Damascus University, Damascus, Syria.
Locations (1):
- Orient Hospital, Damascus, Syria

REFERENCES:
- [Background] Aguilar-Rojas A, Huerta-Reyes M. Human gonadotropin-releasing hormone receptor-activated cellular functions and signaling pathways in extra-pituitary tissues and cancer cells (Review). Oncol Rep. 2009 Nov;22(5):981-90. doi: 10.3892/or_00000525. PMID 19787210
- [Background] Cheung LW, Wong AS. Gonadotropin-releasing hormone: GnRH receptor signaling in extrapituitary tissues. FEBS J. 2008 Nov;275(22):5479-95. doi: 10.1111/j.1742-4658.2008.06677.x. PMID 18959738
- [Background] Setti AS, Figueira RC, de Almeida Ferreira Braga DP, Azevedo MC, Iaconelli A Jr, Borges E Jr. Oocytes with smooth endoplasmic reticulum clusters originate blastocysts with impaired implantation potential. Fertil Steril. 2016 Dec;106(7):1718-1724. doi: 10.1016/j.fertnstert.2016.09.006. Epub 2016 Oct 12. PMID 27743693
- [Background] Sfontouris IA, Lainas GT, Lainas TG, Faros E, Banti M, Kardara K, Anagnostopoulou K, Kontos H, Petsas GK, Kolibianakis EM. Complex chromosomal aberrations in a fetus originating from oocytes with smooth endoplasmic reticulum (SER) aggregates. Syst Biol Reprod Med. 2018 Aug;64(4):283-290. doi: 10.1080/19396368.2018.1466375. Epub 2018 May 2. PMID 29718716
- [Background] Stigliani S, Moretti S, Casciano I, Canepa P, Remorgida V, Anserini P, Scaruffi P. Presence of aggregates of smooth endoplasmic reticulum in MII oocytes affects oocyte competence: molecular-based evidence. Mol Hum Reprod. 2018 Jun 1;24(6):310-317. doi: 10.1093/molehr/gay018. PMID 29635518
- [Background] Setti AS, Figueira RC, Braga DP, Colturato SS, Iaconelli A Jr, Borges E Jr. Relationship between oocyte abnormal morphology and intracytoplasmic sperm injection outcomes: a meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2011 Dec;159(2):364-70. doi: 10.1016/j.ejogrb.2011.07.031. Epub 2011 Aug 6. PMID 21824710
- [Background] Lazzaroni-Tealdi E, Barad DH, Albertini DF, Yu Y, Kushnir VA, Russell H, Wu YG, Gleicher N. Oocyte Scoring Enhances Embryo-Scoring in Predicting Pregnancy Chances with IVF Where It Counts Most. PLoS One. 2015 Dec 2;10(12):e0143632. doi: 10.1371/journal.pone.0143632. eCollection 2015. PMID 26630267
- [Background] Cota AM, Oliveira JB, Petersen CG, Mauri AL, Massaro FC, Silva LF, Nicoletti A, Cavagna M, Baruffi RL, Franco JG Jr. GnRH agonist versus GnRH antagonist in assisted reproduction cycles: oocyte morphology. Reprod Biol Endocrinol. 2012 Apr 27;10:33. doi: 10.1186/1477-7827-10-33. PMID 22540993
- [Background] Zanetti BF, Braga DPAF, Setti AS, Iaconelli A Jr, Borges E Jr. Effect of GnRH analogues for pituitary suppression on oocyte morphology in repeated ovarian stimulation cycles. JBRA Assist Reprod. 2020 Jan 30;24(1):24-29. doi: 10.5935/1518-0557.20190050. PMID 31436072
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182